CLINICAL TRIAL: NCT00000707
Title: Aerosols in the Treatment of Asymptomatic Pneumocystis Pneumonia: A Pilot Study Assessing the Effectiveness of Aerosolized Pentamidine as Treatment of Subclinical Pneumocystis Infection in Patients With No Clinical Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 048; 11022 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Respiratory Function Tests; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Lung; HIV Seropositivity; Drug Evaluation; Administration, Inhalation; Aerosols; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; HIV Seropositivity; Respiratory Aspiration; Acquired Immunodeficiency Syndrome | interventions — Pentamidine

INTERVENTIONS:
Drug: Pentamidine isethionate

SUMMARY:
To confirm the ability of pulmonary (lung) function testing (PFT) to detect Pneumocystis carinii pneumonia (PCP) before the development of clinical symptoms and to determine if pentamidine (PEN), a drug used in treating PCP, can be given effectively as an aerosol (inhaled mist). Other goals include the measurement of the actual amount of PEN that reaches the lung, and to determine if close clinical observation is safer and as effective as drug therapy for the prevention of subsequent episodes of PCP.

Many AIDS patients develop PCP, but the effectiveness of early diagnosis and treatment of PCP is not known. The effectiveness of PEN may be improved if treatment is begun when the parasite burden (the number of organisms in the lung) is still small, and before respiratory symptoms appear. If PFT of HIV-infected patients is able to identify patients in the early stages of infection, outpatient treatment of these patients offers a possible alternative to the expense and toxicity of continuous preventive therapy of all high-risk patients.

DETAILED DESCRIPTION:
Many AIDS patients develop PCP, but the effectiveness of early diagnosis and treatment of PCP is not known. The effectiveness of PEN may be improved if treatment is begun when the parasite burden (the number of organisms in the lung) is still small, and before respiratory symptoms appear. If PFT of HIV-infected patients is able to identify patients in the early stages of infection, outpatient treatment of these patients offers a possible alternative to the expense and toxicity of continuous preventive therapy of all high-risk patients.

Patients are treated with aerosolized PEN on an outpatient basis. The aerosol therapy is given by a respiratory therapist 5 times a week, for a total of 21 days of treatment. In addition, patients participate in two radioactive aerosol studies in which the patient inhales a radioactive gas while sitting with his/her back against a gamma camera. The resulting picture outlines the lungs. Then the gas is exhaled and the patient breathes an aerosol of PEN. This mist contains a single dose of PEN mixed with a small amount of radioactivity (99mTc-pertechnetate). The gamma camera determines where the particles deposit in the lungs. The radioactive exposure is equivalent to a typical x-ray of the ribs. Patients also undergo diagnostic bronchoscopy with lavage, and PFT. Blood is drawn to measure the blood level of PEN. Patients are followed (clinical exams and PFT's) for 6 months after the end of therapy. Prophylaxis for PCP is allowed during the 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria

Concurrent Treatment:

Allowed during aerosolization:

Metaproterenol or albuterol to treat bronchospasm.

Patients must have:

* HIV infection confirmed by ELISA, HIV culture, or p24 antigenemia.
* Suspected subclinical Pneumocystis carinii infection as detected by > 10 percent change in lung volumes and/or diffusing capacity indicative of progressive restrictive disease as detected by monthly screening pulmonary function tests (PFT's). Patients will be afebrile and have no respiratory signs or symptoms of clinical disease. Morphologic confirmation of pneumocysts will be determined by bronchoalveolar lavage (BAL) performed 24 hours after the initial aerosol inhalation. If the BAL is negative for pneumocysts, the patient will be withdrawn from this protocol and will be followed per the screening PFT protocol at Stony Brook.
* Diagnostic bronchoscopy and BAL must be performed within 2 weeks of detection of > 10 percent change in PFTs.
* Ability and willingness to sign informed consent.

Prior Medication:

Allowed:

* Primary prophylaxis with agents active against Pneumocystis carinii pneumonia (PCP), but no more than 5 patients may have received prior prophylaxis with aerosolized pentamidine.
* Zidovudine.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* History of Pneumocystis carinii pneumonia (PCP).
* Development of respiratory signs and/or symptoms in the interval between detection of pulmonary function test (PFT) abnormality and the time of initial aerosol deposition.
* Dyspnea, cough, or bronchospasm that prevents cooperation with aerosol administration.
* History of a major adverse reaction to pentamidine defined by absolute neutropenia, < 750 polymorphonuclear leukocytes plus bands; thrombocytopenia, < 40000 platelets; creatinine rise, > 3.0 mg/dl; liver function abnormalities, SGOT or SGPT > 5 x normal; hypoglycemia, < 50 mg/dl; rash, exfoliative or mucositis; cough, unremitting cough or bronchospasm uncontrolled by bronchodilator preventing > 50 percent of dose delivered for > 2 days.

Concurrent Medication:

Excluded:

* Zidovudine.

Patients unable to cooperate with aerosol administration are excluded.

Prior Medication:

Excluded:

- Another antiprotozoal regimen for this episode. Unable to complete therapy or follow-up for social reasons in the opinion of the investigator.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Study Completion 1991-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Smaldone G, Study Chair
Locations (1):
- SUNY - Stony Brook, Stony Brook, New York, United States

REFERENCES:
- [Background] Smaldone GC, Fuhrer J, Steigbigel RT, McPeck M. Factors determining pulmonary deposition of aerosolized pentamidine in patients with human immunodeficiency virus infection. Am Rev Respir Dis. 1991 Apr;143(4 Pt 1):727-37. doi: 10.1164/ajrccm/143.4_Pt_1.727. PMID 2008984